CLINICAL TRIAL: NCT05406921
Title: Implementation of MIND at Home Program in Primary Care for People Living With Dementia: A Pilot Study
Brief Title: Implementation of MIND at Home Into Primary Care for People Living With Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: American Medical Group Association (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Brown University (Other); Johns Hopkins University (Other); McFarland Clinic (Unknown); Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: FY21_Pilot1_Ciemins; 3U54AG063546-03 (NIH)
Record Dates: First submitted 2022-06-01; First posted 2022-06-07 (Actual); Results first posted 2025-01-31 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Dementia
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention Arm: PLWD (Experimental): 100 community-residing PC patients with an ADRD diagnosis will be enrolled and receive MIND coordination services for 3 months to test program implementation feasibility in PC practice settings.
  Interventions: Behavioral: MIND at Home
- Data Validation Arm (No Intervention): An additional 100 PLWD will serve as a data validation arm to demonstrate the feasibility of collecting and validating data from large health systems.
- Intervention Arm: PLWD CPs (Experimental): 100 Care Partners (CPs) of the 100 community-residing PC patients with an ADRD diagnosis will be enrolled and receive MIND coordination services for 3 months to test program implementation feasibility in PC practice settings.
  Interventions: Behavioral: MIND at Home

INTERVENTIONS:
Behavioral: MIND at Home — Maximizing Independence at Home-MIND at Home (MIND) is a comprehensive care coordination program born from geriatric psychiatry. This model takes an interdisciplinary, collaborative care approach to care by systematically assessing and addressing a wide range of dementia-care related needs of both PLWD and their care partners that place both at increased risk for poor outcomes.
  Arms: Intervention Arm: PLWD; Intervention Arm: PLWD CPs

SUMMARY:
The number of people living with dementia (PLWD) is growing. PLWD are often cared for at home by an informal caregiver, but this care is often not sufficient, resulting in costly hospitalizations and other unnecessary and avoidable use of health services. In addition, many PLWD are transferred to costly long-term care facilities despite their preference to live at home. One way to improve care for PLWD is to work with their primary care doctors to provide better quality of care at lower costs for their patients. To accomplish this, we propose to collaboratively implement the MIND at Home Dementia Care Coordination Program into primary care clinics. The program expands the skills of existing primary care staff to the level of Memory Care Coordinators (MCCs), who will work with a larger primary care team on combining the benefits of clinic-based services with home-based services that support PLWD, their families, and care partners.

Two health care organizations will enroll 150 people in the MIND at Home program for 3 months at a time. The program includes one home visit per month, a comprehensive needs assessment (which assesses medical, nonmedical, social, and environmental issues), the subsequent development and implementation of an individualized care plan, and unlimited contact with the MCC for the PLWD, their family, and care partner. The primary care team, including the MCC, will also have access to weekly virtual sessions focused on dementia and including short lectures and the discussion of specific case examples.

Rates of monthly hospitalizations among participants and emergency room (ER) visits and number of medications the PLWD takes every month will be collected from the health care organization. The hypothesis is that the rate of hospitalizations and ER visits will decrease, and the number of medications will also decrease. We hope to positively impact the quality and costs of care associated with caring for PLWD.

This pilot seeks to test the feasibility of implementing the MIND at Home program into primary care in a racially, ethnically, and geographically diverse population of PLWD to prepare for a larger study that will determine this program's effectiveness and spread it broadly into primary care clinics across the country.

From the perspectives of health systems and overall society, MIND at Home will reduce costs, improve primary care team satisfaction, and preserve the dignity and independence of PLWD by enabling them to age at home.

DETAILED DESCRIPTION:
Integration of evidence-based collaborative care management models such as the MIND at Home Dementia Care Coordination Program within Primary Care (PC) aligns with the Centers for Medicare and Medicaid Services (CMS) initiatives to provide advanced PC services to an especially complex and costly patient group and aligns with AHRQ's team-based Collaborative Care Model. This project will embed and test the feasibility of a novel best practice-based approach, MIND at Home, within PC to enhance and elevate the role of existing PC staff to Memory Care Coordinators (MCCs), increase PC access to interdisciplinary collaborative care, and systematically combines the benefits of clinic-based services with home-based assessment to support family-centered care planning and implementation for PLWD and their care partners. Weekly virtual collaborative learning sessions that include geriatric psychiatry consultants augment the PC care team's work to support the development and mastery of dementia assessment and care management skills and confidence at the PC sites. Our overarching goal is to test and establish feasibility, acceptability, fidelity, and sample size/referral rate data for MIND at Home in PC to prepare for a future multi-site embedded pragmatic trial.

Aim 1: Evaluate the feasibility and validity of eligible PLWD identification, referral, and enrollment in a best practice-based dementia care coordination program (MIND at Home) at 3 primary care clinics. Algorithms based on CMS's Chronic Care Warehouse definition of Alzheimer's Disease (AD) or AD and Related Dementias (ADRD) will be deployed in each respective clinic's electronic health record (EHR) to identify eligible PLWD and standardized referral and enrollment protocols will be enacted. Referral, recruitment, patient acceptance, and attrition rates will be calculated to assess the feasibility of use of the algorithm and of the recruitment protocol. Health equity in recruitment and enrollment will be assessed by comparing demographics (race/ethnicity) of program enrollees with the background population e.g., clinic ADRD patient panel, and by comparing enrollment of rural vs. suburban PC sites.

Aim 2: Evaluate the feasibility, acceptability, and fidelity of implementing MIND at Home in 3 primary care clinics in 2 geographically and demographically diverse integrated health systems. Using a pragmatic trial design, 150 community-residing PC patients with an ADRD diagnosis will be enrolled, each for a 3-month period. Program enrollees will receive office- plus home-based dementia care assessment, individualized care planning, and implementation by an interdisciplinary PC-based team, supported by regular case-based learning sessions. Implementation will be assessed by collecting a standard set of delivery workflow process, clinical, and health care utilization metrics. The investigators will assess feasibility through referral, enrollment, and retention rates, number of MCC-dyad contacts, and clinic staff participation in weekly tele-collaboratives. Fidelity will be assessed through tracking the completion of intervention components and PC team self-evaluation. The investigators will survey clinic staff on perceived program acceptability, usefulness, and challenges/unintended consequences. Program implementation will be tailored to accommodate diverse dyads (PLWD + care partner), which will be closely monitored and tracked.

Aim 3: Evaluate the feasibility of ascertainment of patient-level outcomes over time using electronic health record (EHR) data. The primary outcome (hospital transfers including admissions, ER visits, and observation stays without admissions), and secondary outcomes (number of medications for enrolled patients) will be gathered using EHR data. Accuracy of ascertainment will be tested through chart review. All clinical outcomes will be collected as time-stamped events for each enrolled patient retrospectively for 3 months prior to enrollment, during enrollment (3 months), and 1-month post-enrollment (total observation=7 months). All outcomes will be assessed by race, ethnicity, and rurality of the PLWD.

Embedding a collaborative, best-practice-based approach such as MIND at Home into PC is a potentially powerful strategy to organize care, improve quality, reduce costs, and maximize the population-level benefit for PLWD. This proposal tests the feasibility of implementing MIND at Home into PC in a racially, ethnically, and geographically diverse PLWD population in order to prepare for a multisite embedded pragmatic clinical trial (ePCT) to evaluate effectiveness, and eventually support broader dissemination and uptake in PC.

ELIGIBILITY:
Inclusion Criteria:

* Community residing adults, ≥18 years
* People Living with Dementia (PLWD) defined by a diagnosis using algorithms based on CMS' Chronic Care Warehouse definition of Alzheimer's Disease, Related Dementias, Related Disorders, and Senile Dementia.11 This definition includes those who have an eligible diagnosis code on any eligible claim (i.e., inpatient, outpatient, skilled nursing facility (SNF), or home health visit or stay) in the past three years or a diagnosis on the patient problem list.
* Actively receiving primary care services at one of three primary care practices within two participating health care organizations selected as study sites.
* Have a reliable care partner who speaks English (or a language spoken by the Memory Care Coordinator).
* Willing to participate in all study home visits and related activities for the entire length of the study (3 months).

Exclusion Criteria:

* PLWD in crisis, e.g., show signs of abuse, neglect, extreme risk of danger to self or others), will be connected to appropriate services, but will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 410 (Actual)
Dates: Start 2022-07-18 (Actual); Primary Completion 2024-04-05 (Actual); Study Completion 2024-06-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth L Ciemins, PhD, Principal Investigator — American Medical Group Association
Locations (2):
- United States (2):
  - McFarland Clinic, Ames, Iowa
  - Atrium Health Wake Forest Baptist Medical Center, Winston-Salem, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Olsen C, Pedersen I, Bergland A, Enders-Slegers MJ, Joranson N, Calogiuri G, Ihlebaek C. Differences in quality of life in home-dwelling persons and nursing home residents with dementia - a cross-sectional study. BMC Geriatr. 2016 Jul 11;16:137. doi: 10.1186/s12877-016-0312-4. PMID 27400744
- [Background] Samus QM, Johnston D, Black BS, Hess E, Lyman C, Vavilikolanu A, Pollutra J, Leoutsakos JM, Gitlin LN, Rabins PV, Lyketsos CG. A multidimensional home-based care coordination intervention for elders with memory disorders: the maximizing independence at home (MIND) pilot randomized trial. Am J Geriatr Psychiatry. 2014 Apr;22(4):398-414. doi: 10.1016/j.jagp.2013.12.175. Epub 2014 Jan 4. PMID 24502822
- [Background] Tanner JA, Black BS, Johnston D, Hess E, Leoutsakos JM, Gitlin LN, Rabins PV, Lyketsos CG, Samus QM. A randomized controlled trial of a community-based dementia care coordination intervention: effects of MIND at Home on caregiver outcomes. Am J Geriatr Psychiatry. 2015 Apr;23(4):391-402. doi: 10.1016/j.jagp.2014.08.002. Epub 2014 Aug 13. PMID 25260557
- [Background] Samus QM, Black BS, Reuland M, Leoutsakos JS, Pizzi L, Frick KD, Roth DL, Gitlin LN, Lyketsos CG, Johnston D. MIND at Home-Streamlined: Study protocol for a randomized trial of home-based care coordination for persons with dementia and their caregivers. Contemp Clin Trials. 2018 Aug;71:103-112. doi: 10.1016/j.cct.2018.05.009. Epub 2018 May 18. PMID 29783091
- [Background] Samus QM, Davis K, Willink A, Black BS, Reuland M, Leoutsakos J, Roth DL, Wolff J, Gitlin LN, Lyketsos CG, Johnston D. Comprehensive home-based care coordination for vulnerable elders with dementia: Maximizing Independence at Home-Plus-Study protocol. Int J Care Coord. 2017 Dec;20(4):123-134. doi: 10.1177/2053434517744071. Epub 2017 Dec 14. PMID 29607051
- [Background] Black BS, Johnston D, Leoutsakos J, Reuland M, Kelly J, Amjad H, Davis K, Willink A, Sloan D, Lyketsos C, Samus QM. Unmet needs in community-living persons with dementia are common, often non-medical and related to patient and caregiver characteristics. Int Psychogeriatr. 2019 Nov;31(11):1643-1654. doi: 10.1017/S1041610218002296. Epub 2019 Feb 4. PMID 30714564
- [Background] Black BS, Johnston D, Rabins PV, Morrison A, Lyketsos C, Samus QM. Unmet needs of community-residing persons with dementia and their informal caregivers: findings from the maximizing independence at home study. J Am Geriatr Soc. 2013 Dec;61(12):2087-2095. doi: 10.1111/jgs.12549. PMID 24479141
- [Background] Hughes TB, Black BS, Albert M, Gitlin LN, Johnson DM, Lyketsos CG, Samus QM. Correlates of objective and subjective measures of caregiver burden among dementia caregivers: influence of unmet patient and caregiver dementia-related care needs. Int Psychogeriatr. 2014 Nov;26(11):1875-83. doi: 10.1017/S1041610214001240. Epub 2014 Aug 8. PMID 25104063
- [Background] Willink A, Davis K, Johnston DM, Black B, Reuland M, Stockwell I, Amjad H, Lyketsos CG, Samus QM. Cost-Effective Care Coordination for People With Dementia at Home. Innov Aging. 2020 Jan 1;4(2):igz051. doi: 10.1093/geroni/igz051. eCollection 2020. PMID 31911954
- [Background] Amjad H, Roth DL, Samus QM, Yasar S, Wolff JL. Potentially Unsafe Activities and Living Conditions of Older Adults with Dementia. J Am Geriatr Soc. 2016 Jun;64(6):1223-32. doi: 10.1111/jgs.14164. Epub 2016 Jun 2. PMID 27253366
- [Background] Taylor DH Jr, Fillenbaum GG, Ezell ME. The accuracy of medicare claims data in identifying Alzheimer's disease. J Clin Epidemiol. 2002 Sep;55(9):929-37. doi: 10.1016/s0895-4356(02)00452-3. PMID 12393082

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention Arm: PLWD: 105 community-residing PC patients with an ADRD diagnosis were enrolled and received MIND coordination services for 3 months to test program implementation feasibility in PC practice settings.
  MIND at Home: Maximizing Independence at Home-MIND at Home (MIND) is a comprehensive care coordination program born from geriatric psychiatry. This model takes an interdisciplinary, collaborative care approach to care by systematically assessing and addressing a wide range of dementia care related needs of both PLWD and their care partners that place both at increased risk for poor outcomes.
- Data Validation Arm: An additional 200 PLWD served as a data validation arm to demonstrate the feasibility of collecting and validating data from large health systems.
- Intervention Arm: PLWD CPs: 105 Care Partners (CPs) of the 105 community-residing PC patients with an ADRD diagnosis were enrolled and received MIND coordination services for 3 months to test program implementation feasibility in PC practice settings.
  MIND at Home: Maximizing Independence at Home-MIND at Home (MIND) is a comprehensive care coordination program born from geriatric psychiatry. This model takes an interdisciplinary, collaborative care approach to care by systematically assessing and addressing a wide range of dementia care related needs of both PLWD and their care partners that place both at increased risk for poor outcomes.
Period: Overall Study
Arm/Group | Intervention Arm: PLWD | Data Validation Arm | Intervention Arm: PLWD CPs
Started | 105 | 200 | 105
Completed | 80 | 188 | 80
Not Completed | 25 | 12 | 25
Not completed — Withdrawal by Subject | 25 | 0 | 25
Not completed — Protocol Violation | 0 | 12 | 0

BASELINE CHARACTERISTICS:
Population: Analysis was conducted on intervention and data validation patients only and per-protocol.
Groups:
- Intervention Arm: PLWD: 105 community-residing PC patients with an ADRD diagnosis were enrolled and received MIND coordination services for 3 months to test program implementation feasibility in PC practice settings.
  MIND at Home: Maximizing Independence at Home-MIND at Home (MIND) is a comprehensive care coordination program born from geriatric psychiatry. This model takes an interdisciplinary, collaborative care approach to care by systematically assessing and addressing a wide range of dementia-care related needs of both PLWD and their care partners that place both at increased risk for poor outcomes.
- Intervention Arm: PLWD CPs: 105 Care Partners (CPs) of the 105 community-residing PC patients with an ADRD diagnosis were enrolled and received MIND coordination services for 3 months to test program implementation feasibility in PC practice settings.
  MIND at Home: Maximizing Independence at Home-MIND at Home (MIND) is a comprehensive care coordination program born from geriatric psychiatry. This model takes an interdisciplinary, collaborative care approach to care by systematically assessing and addressing a wide range of dementia-care related needs of both PLWD and their care partners that place both at increased risk for poor outcomes.
- Total: Total of all reporting groups
Arm/Group | Intervention Arm: PLWD | Data Validation Arm | Intervention Arm: PLWD CPs | Total
Number analyzed (Participants) | 80 | 188 | 80 | 348
Age, Continuous [Mean (Standard Deviation); unit: years] | 81 (6.18) | 79 (9.16) | NA (NA) — We did not collect age of Care Partners. | 80 (7.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 96 | 53 | 188
  Male | 41 | 92 | 27 | 160
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 1 | 6
  Not Hispanic or Latino | 77 | 183 | 79 | 339
  Unknown or Not Reported | 1 | 2 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 9 | 25 | 9 | 43
  White | 69 | 158 | 70 | 297
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 5 | 0 | 6
Region of Enrollment [Number; unit: participants]
  United States | 80 | 188 | 80 | 348
hospital transfers [Mean (Standard Deviation); unit: hospital transfers per 1000 person days] | 1.89 (5.78) | 2.50 (8.29) | NA (NA) — We did not collect encounter day on the care partners. | 2.07 (6.62)

OUTCOME MEASURES:

1. Primary Outcome: Change in Number of Hospital Transfers Pre/Post Intervention
Description: Hospital transfers include hospitalizations, emergency department visits, and observation stays without admission.
Time Frame: Data will be collected monthly for the 3 months prior to enrollment, the 3 months during enrollment, and one month post enrollment.
Population: Per-protocol analysis.
Measure: Mean (Standard Deviation); unit: hospital transfers per 1000 person days
Arm/Group | Intervention Arm: PLWD | Data Validation Arm | Intervention Arm: PLWD CPs
Number analyzed (Participants) | 80 | 188 | 80
hospital transfers per 1000 person days | 0.97 (7.94) | 0.65 (7.10) | NA (NA) — We did not collect outcomes on CPs.

2. Secondary Outcome: Change in Number of Medications Pre/Post Intervention
Description: The secondary outcomes are number of total medications, number of anti-psychotics, acetylcholinesterase inhibitors, and memantine medications.
Time Frame: as for outcome 1
Population: Only one site was able to provide data on total medications.
Measure: Mean (Standard Deviation); unit: number of medications
Arm/Group | Intervention Arm: PLWD | Data Validation Arm | Intervention Arm: PLWD CPs
Number analyzed (Participants) | 46 | 100 | 46
number of medications | -0.43 (3.99) | 0.33 (2.44) | NA (NA) — We did not collect outcome data on CPs.
Statistical Analysis 1: Comparison: Data Validation Arm; This was a feasibility study and not powered to detect significant differences pre-/post-intervention; Test type: Superiority; p < 0.05, ANOVA; Mean Difference (Net) = 0.32

ADVERSE EVENTS:
Time Frame: Adverse event data were collected on each intervention patient from date of study enrollment through the conclusion of the 3-month study period.
Description: We did not collect AEs on Care Partners nor were we able to given that they were not necessarily patients of the same health systems with which we partnered.
  We did not collect AEs on patients in the data validation arm as we had no contact with those patients.
  In both of these groups, All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Groups:
- Intervention Arm: PLWD: 80 community-residing PC patients with an ADRD diagnosis were enrolled and received MIND coordination services for 3 months to test program implementation feasibility in PC practice settings.
  MIND at Home: Maximizing Independence at Home-MIND at Home (MIND) is a comprehensive care coordination program born from geriatric psychiatry. This model takes an interdisciplinary, collaborative care approach to care by systematically assessing and addressing a wide range of dementia-care related needs of both PLWD and their care partners that place both at increased risk for poor outcomes.
- Data Validation Arm: An additional 188 PLWD served as a data validation arm to demonstrate the feasibility of collecting and validating data from large health systems.
- Intervention Arm: PLWD CPs: 80 Care Partners (CPs) of the 105 community-residing PC patients with an ADRD diagnosis were enrolled and received MIND coordination services for 3 months to test program implementation feasibility in PC practice settings.
  MIND at Home: Maximizing Independence at Home-MIND at Home (MIND) is a comprehensive care coordination program born from geriatric psychiatry. This model takes an interdisciplinary, collaborative care approach to care by systematically assessing and addressing a wide range of dementia-care related needs of both PLWD and their care partners that place both at increased risk for poor outcomes.
Arm/Group | Intervention Arm: PLWD | Data Validation Arm | Intervention Arm: PLWD CPs
All-Cause Mortality (participants affected / at risk) | 2/105 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 29/105 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/105 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention Arm: PLWD (N=105) | Data Validation Arm (N=0) | Intervention Arm: PLWD CPs (N=0)
Hospitalization (Injury, poisoning and procedural complications) | 7 (7) | NA | NA
Hospitalization (Cardiac disorders) | 1 (1) | NA | NA
Hospitalization (Respiratory, thoracic and mediastinal disorders) | 7 (7) | NA | NA
Change in level of care (Nervous system disorders) | 5 (5) | NA | NA
Hospitalization (Investigations) | 1 (1) | NA | NA
ED Visit (Nervous system disorders) | 3 (6) | NA | NA
Changed Level of Care (Social circumstances) | 1 (1) | NA | NA
ED Visit (Injury, poisoning and procedural complications) | 2 (2) | NA | NA
ED Visit (Gastrointestinal disorders) | 2 (2) | NA | NA

LIMITATIONS AND CAVEATS:
This was designed as a pilot feasibility study. The intent was to determine the feasibility of (1) implementing the program in primary care, and (2) collecting patient-level data from health systems. Therefore it was not powered to find statistically significant results, although we still conducted an analysis and submitted results. Per our protocol, we collected only minimal data on Care Partners. They were not always patients of the same health system as the PLWD.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-07-25): https://cdn.clinicaltrials.gov/large-docs/21/NCT05406921/Prot_SAP_000.pdf